CLINICAL TRIAL: NCT05648279
Title: Personalized Hemodynamic Management Targeting Preoperative Baseline Cardiac Index in High-risk Patients Having Major Abdominal Surgery: the International Multicenter Randomized PELICAN Trial
Brief Title: Personalized Hemodynamic Management in High-risk Major Abdominal Surgery
Acronym: PELICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-100955-BO-ff
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Output; Surgery; Postoperative Complications; Anesthesia
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In patients in the routine management group, the treating anesthesiologists will be blinded to data of preoperative baseline cardiac output measurements to avoid performance bias. Participanting patients, outcome assessors, and data analysts are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine hemodynamic management (control) (No Intervention): In patients assigned to routine hemodynamic management, hemodynamic management will performed as per anesthesiologist preference. Cardiac index monitoring will be will measured using the Baxter Starling Fluid Management System (Baxter, Deerfield, IL, USA). The attending anesthesiologist will be blinded to cardiac index measurements. Cardiac index monitoring can be unblinded upon request. Mean arterial blood pressure will be maintained above 65 mmHg.
- Personalized hemodynamic management (intervention) (Experimental): In patients assigned to personalized hemodynamic management, intraoperative cardiac index will be maintained at least at the preoperative baseline cardiac index using a predefined treatment algorithm.
  Preoperative baseline cardiac index will be determined with the patient being awake and resting in supine position using the Starling Fluid Management System (Baxter, Deerfield, IL, USA) (usually at least one day before surgery). We will define the individual preoperative baseline cardiac index as the average value over a 5 min period at rest (minimum cardiac index threshold: 2.2 L min-1 m-2).
  Mean arterial blood pressure will be maintained above 65 mmHg. The study intervention will start at the beginning of surgery and will end at the end of surgery.
  Interventions: Other: Personalized hemodynamic management

INTERVENTIONS:
Other: Personalized hemodynamic management — Personalized hemodynamic management: Intraoperative cardiac index will be maintained at least at the preoperative baseline cardiac index. Preoperative baseline cardiac index will be determined one day before surgery with the patient being awake and resting in the supine position using the Starling Fluid Management System (Baxter, Deerfield, IL, USA) Preoperative baseline cardiac index will be determined with the patient being awake and resting in supine position using the Starling Fluid Management System (Baxter, Deerfield, IL, USA) (usually at least one day before surgery). We will define the individual preoperative baseline cardiac index as the average value over a 5 min period at rest (minimum cardiac index threshold: 2.2 L min-1 m-2). Intraoperative cardiac index will be measured using the Baxter Starling Fluid Management System.
  Arms: Personalized hemodynamic management (intervention)

SUMMARY:
Postoperative mortality within 30 days after surgery is around 2% in patients having major noncardiac surgery in Europe and the USA. In fact, if the first 30 days after surgery were considered a disease, it would be the third leading cause of death globally. Postoperative deaths are a consequence of postoperative organ injury and complications - including acute myocardial injury, acute kidney injury, and severe infectious complications. To avoid postoperative deaths, it is thus crucial to reduce postoperative organ injury and complications. To reduce postoperative organ injury and complications, modifiable risk factors need to be addressed. These modifiable risk factors for postoperative organ injury include low blood flow states and intraoperative hypotension. Optimizing blood flow (i.e., cardiac index) during surgery may thus be effective in reducing postoperative organ injury and complications. However, the optimal hemodynamic treatment strategy for high-risk surgical patients remains unclear. Cardiac index varies substantially between individuals. However, current intraoperative hemodynamic treatment strategies mainly aim to maximize cardiac index instead of using personalized cardiac index targets for each individual patient. A single-center pilot trial suggests that using individualized cardiac index targets during surgery may reduce postoperative organ injury and complications compared to routine hemodynamic management. However, large robust trials investigating the effect of personalized hemodynamic management targeting preoperative baseline cardiac index on postoperative complications are missing.

The investigators, therefore, propose a multicenter randomized trial to test the hypothesis that personalized intraoperative hemodynamic management targeting preoperative baseline cardiac index reduces the incidence of a composite outcome of acute kidney injury, acute myocardial injury, non-fatal cardiac arrest, severe infectious complications, and death within 7 days after surgery compared to routine hemodynamic management in high-risk patients having elective major abdominal surgery.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

Consenting patients ≥45 years scheduled for elective major abdominal surgery (involving visceral organs) under general anesthesia that is expected to last ≥90 minutes AND presence of ≥1 of the following high-risk criteria:

* exercise tolerance <4 metabolic equivalents as defined by the guidelines of the American College of Cardiology/American Heart Association
* renal impairment (serum creatinine ≥1.3 mg dL-1 or estimated glomerular filtration rate <90 mL min-1 (1.73 m2)-1 within the last 6 months
* coronary artery disease
* chronic heart failure (New York Heart Association Functional Classification ≥II)
* valvular heart disease (moderate or severe)
* history of stroke
* peripheral arterial occlusive disease (any stage)
* chronic obstructive pulmonary disease (any stage) or pulmonary fibrosis (any stage)
* diabetes mellitus requiring oral hypoglycemic agent or insulin
* immunodeficiency due to a disease (e.g., HIV, leukemia, multiple myeloma) or therapy (e.g., immunosuppressants, chemotherapy, radiation, steroids [above Cushing threshold])
* liver cirrhosis (any Child-Pugh class)
* body mass index ≥30 kg m-2
* history of smoking within two years of surgery
* age ≥65 years
* expected surgery duration ≥180 minutes
* B-type natriuretic peptide (BNP) >80 ng/L or N-terminal B-type natriuretic peptide (NT-proBNP) >200 ng/L within the last 6 months

Exclusion Criteria:

* emergency surgery
* ambulatory surgery
* planned surgery: nephrectomy, liver or kidney transplantation surgery
* status post transplantation of kidney, liver, heart, or lung
* sepsis (according to current Sepsis-3 definition)
* American Society of Anesthesiologists physical status classification V or VI
* pregnancy
* impossibility to perform cardiac index monitoring using the Starling Fluid Management System (Baxter, Deerfield, IL, USA)
* current participation in another clinical trial or treatment with a similar biological mechanism or primary outcome measure

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-10-25 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Composite outcome of major postoperative complications | Postoperative Day 7
  Collapsed composite ("any event versus none") of acute kidney injury, acute myocardial injury (including myocardial infarction), non-fatal cardiac arrest, severe infectious complications, and death within 7 days after surgery.

SECONDARY OUTCOMES:
Composite outcome of major postoperative complications | Postoperative Day 3
  Collapsed incidence of acute kidney injury, acute myocardial injury (including myocardial infarction), non-fatal cardiac arrest, severe infectious complications, and death within 3 days after surgery.
Postoperative acute kidney injury | Postoperative Day 3
  Incidence of acute kidney injury within 3 days after surgery
Postoperative acute kidney injury | Postoperative Day 7
  Incidence of acute kidney injury within 7 days after surgery
Postoperative acute myocardial injury | Postoperative Day 3
  Incidence of acute myocardial injury within 3 days after surgery
Postoperative acute myocardial injury | Postoperative Day 7
  Incidence of acute myocardial injury within 7 days after surgery
Postoperative severe infectious complications | Postoperative Day 3
  Incidence of a composite outcome of fever, respiratory infection, neurological infection, urinary system infection, colitis or infection with Clostridium difficile, endometritis, surgical site infection, deep incisional surgical site infection, organ or space surgical site infection (including anastomotic leak), unknown infection with pathogenic organisms in tissue or fluid, and sepsis within 3 days after surgery.
Postoperative severe infectious complications | Postoperative Day 7
  Incidence of a composite outcome of fever, respiratory infection, neurological infection, urinary system infection, colitis or infection with Clostridium difficile, endometritis, surgical site infection, deep incisional surgical site infection, organ or space surgical site infection (including anastomotic leak), unknown infection with pathogenic organisms in tissue or fluid, and sepsis within 7 days after surgery.
Postoperative non-fatal cardiac arrest | Postoperative Day 3
  Incidence of postoperative non-fatal cardiac arrest within 3 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 7
  Incidence of postoperative non-fatal cardiac arrest within 7 days after surgery
Postoperative death | Postoperative Day 3
  Incidence of postoperative death within 3 days after surgery
Postoperative death | Postoperative Day 7
  Incidence of postoperative death within 7 days after surgery
Composite outcome of long-term postoperative complications | Postoperative Day 30
  Collapsed incidence of need for renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, and death within 30 days after surgery
Composite outcome of long-term postoperative complications | Postoperative Day 90
  Collapsed incidence of need for renal replacement therapy, myocardial infarction, non-fatal cardiac arrest, and death within 90 days after surgery
Postoperative need for renal replacement therapy | Postoperative Day 30
  Incidence of need for renal replacement therapy within 30 days after surgery
Postoperative need for renal replacement therapy | Postoperative Day 90
  Incidence of need for renal replacement therapy within 90 days after surgery
Postoperative myocardial infarction | Postoperative Day 30
  Incidence of myocardial infarction within 30 days after surgery
Postoperative myocardial infarction | Postoperative Day 90
  Incidence of myocardial infarction within 90 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 30
  Incidence of non-fatal cardiac arrest within 30 days after surgery
Postoperative non-fatal cardiac arrest | Postoperative Day 90
  Incidence of non-fatal cardiac arrest within 90 days after surgery
Postoperative death | Postoperative Day 30
  Incidence of death within 30 days after surgery
Postoperative death | Postoperative Day 90
  Incidence of death within 90 days after surgery
Postoperative fever | Postoperative Day 7
  Incidence of fever within 7 days after surgery
Postoperative respiratory infection | Postoperative Day 7
  Incidence of respiratory infection within 7 days after surgery
Postoperative neurological infection | Postoperative Day 7
  Incidence of neurological infection within 7 days after surgery
Postoperative urinary system infection | Postoperative Day 7
  Incidence of urinary system infection within 7 days after surgery
Postoperative colitis or infection with Clostridium difficile | Postoperative Day 7
  Incidence of colitis or infection with Clostridium difficile within 7 days after surgery
Postoperative endometritis | Postoperative Day 7
  Incidence of endometritis within 7 days after surgery
Postoperative deep incisional surgical site infection | Postoperative Day 7
  Incidence of deep incisional surgical site infection within 7 days after surgery
Postoperative organ or space surgical site infection | Postoperative Day 7
  Incidence of organ or space surgical site infection (including anastomotic leak) within 7 days after surgery
Postoperative unknown infection with pathogenic organisms in tissue or fluid | Postoperative Day 7
  Incidence of unknown infection with pathogenic organisms in tissue or fluid within 7 days after surgery
Postoperative sepsis | Postoperative Day 7
  Incidence of sepsis within 7 days after surgery
Transfer from intensive care unit to normal ward | Postoperative Day 90
  Time-to-event endpoint with the event "transfer from intensive care unit to normal ward" within 90 days after surgery
Hospital discharge | Postoperative Day 90
  Time-to-event endpoint with the event "hospital discharge" within 90 days after surgery
Unplanned hospital re-admission | Postoperative Day 30
  Incidence of unplanned hospital re-admission within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Saugel, M.D., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (12):
- Medical University of Graz, Graz, Austria
- University Hospital Plzen, Pilsen, Czechia
- Denmark (3):
  - Hvidovre Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - University Medical Center Copenhagen Bispebjerg and Frederiksberg, Copenhagen
- Germany (6):
  - University Hospital RWTH Aachen, Aachen
  - University Hospital Düsseldorf, Düsseldorf
  - University Medical Center Hamburg, Hamburg
  - University Medical Center Schleswig Holstein, Lübeck, Lübeck
  - University Hospital Marburg, Marburg
  - LMU Munich, Munich
- Clínica Universidad de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start date 12 months after article publication End date: 5 years after article publication
Access Criteria: Written request to Principal Investigator